CLINICAL TRIAL: NCT06076603
Title: Comparison of Epithelial Lining Fluid and Blood Pharmacokinetics and Pharmacodynamics of Intravenous and Intravenous Plus Nebulized Polymyxin B in Multidrug Resistant Bacteria Ventilator-associated Pneumonia Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jianfeng Xie, MD.PhD, Southeast University, China
Other Study IDs: PMBPIN
Record Dates: First submitted 2023-09-19; First posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Polymyxin B; Ventilator-associated Pneumonia; Multidrug Resistant Bacterial Infection; Pharmacogenomic Drug Interaction
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intravenous combined with nebulized polymyxin B: The intravenous combined nebulization patient group was divided into two subgroups based on the different doses received -25mg q12h and 50mg q12h. Patients in the intravenous combination nebulized polymyxin B group received a total medication dose of 1.25 to 1.5mg/kg, of which 25-50mg was used for nebulization and the remaining portion was used for intravenous administration. The specific method of nebulization is to receive nebulized bronchodilator 30 minutes before nebulization, add 25-50mg of polymyxin B to 5ml of physiological saline for dilution, use a vibrating mesh nebulizer to connect to the patient's ventilator pipeline suction tube, do not change the original ventilator parameter settings, and continue nebulization for 30 minutes. After 30 minutes, regardless of whether there is any residue of the nebulized drug, it will be discarded according to general nursing methods.
  Interventions: Drug: nebulized polymyxin B
- Intravenous polymyxin group B: This group of patients received intravenous injection of polymyxin B alone, with intravenous doses of 1.25-1.5mg/kg of polymyxin B administered every 12 hours.

INTERVENTIONS:
Drug: nebulized polymyxin B — The experimental group received intravenous combined nebulization of polymyxin B
  Groups: Intravenous combined with nebulized polymyxin B

SUMMARY:
The goal of this observational study is to investigate whether intravenous polymyxin B combined with nebulisation achieves better antimicrobial efficacy and clinical outcomes than intravenous use alone in patients with multidrug-resistant gram-negative bacilli infected with ventilator-associated pneumonia. The main questions it aims to answer are:

* When using intravenous polymyxin B to treat patients with ventilator-associated pneumonia caused by multidrug-resistant bacteria in clinical practice, is it necessary to assist with polymyxin B nebulization therapy？
* If necessary, how much dose of nebulization is better? Participants will be divided into two groups based on whether they have received nebulization treatment with polymyxin B in clinical practice. Blood and alveolar lavage fluid samples will be collected after the first dose injection and reaching the steady-state dose, and the drug concentration differences in blood and ELF will be measured in patients who have received intravenous injection of polymyxin B alone and those who have received adjuvant nebulization of polymyxin B, as well as differences in clinical outcomes and side effects.

Researchers will compare the differences in blood and ELF drug concentrations, clinical outcomes, and incidence of side effects between two groups of patients, to see if is it necessary to assist with polymyxin B nebulization therapy in patients with multidrug-resistant gram-negative bacilli infected with ventilator-associated pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years old;
* ICU patients;
* Patients with MDR-infected VAP were diagnosed by etiological culture results;
* Expect to receive at least 6 doses (3 days) of polymyxin B;
* Obtain informed consent;

Exclusion Criteria:

* The patient has a history of severe hypersensitivity to polymyxin B;
* Patients cannot tolerate alveolar lavage;
* Oncology patients,includes hematologic malignancies;
* Pregnant or lactating women;
* Patients with other conditions that the investigators consider unsuitable for enrollment;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Screening of patients with multiple drug-resistant bacterial infections and ventilator-associated pneumonia admitted to the Intensive Care Department of Affiliated Zhongda Hospital of Southeast University. Based on the medical decisions of clinical physicians, they received intravenous administration of polymyxin B alone and intravenous combination nebulization of polymyxin B. Patients were divided into two groups according to the actual treatment methods of polymyxin B.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Blood concentration | 3 days after the end of the patient's first medication use
  Blood concentration
ELF concentration | 3 days after the end of the patient's first medication use
  Drug concentration in ELF solution

SECONDARY OUTCOMES:
28-day clinical cure rate | 28 days after the end of the patient's medication
  the proportion of subjects who are thought as clinical effectiveness 28 days after treatment with polymyxin B to the number of subjects in each group.
28-day microbiological cure rate | 28 days after the end of the patient's medication
  the proportion of subjects of microbiological cure to the number of subjects in each group 28 days after treatment with polymyxin B.
28-day adverse reaction rate | 28 days after the end of the patient's medication
  the proportion of subjects who experienced adverse reactions within 28 days after treatment with polymyxin B to the number of subjects in each group

CONTACTS AND LOCATIONS:
Overall Officials: Yingzi Huang, MD, Study Chair — Department of Critical Care Medicine, Zhongda Hospital, School of Medicine, Southeast University
Locations (1):
- Zhongda Hospital Affiliated to Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No